CLINICAL TRIAL: NCT06842329
Title: "The Effectiveness of Helfer Skin Tap Technique and ShotBlocker in Reducing Pain Severity During Intramuscular Injections in Adolescent Dysmenorrhea: A Randomized Controlled Trial"
Brief Title: The Effect of Distraction Techniques Used in Intramuscular (IM) Injections on Pain in Adolescents Presenting to the Emergency Department With Dysmenorrhea: A Randomized Controlled Study
Acronym: "HSTT-SB Dysme
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu MEZDE (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Sponsor-Investigator, Duygu MEZDE, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-26521195-604.01-256976619; not yet assignet (Other: university of Ondokuz Mayıs)
Record Dates: First submitted 2025-01-31; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Dysmenorrhea; Pain; Distraction Methods
Keywords: helfer skin tap; shotblocker; pain management
MeSH Terms: conditions — Dysmenorrhea; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with a parallel assignment design. Participants will be randomly assigned to one of three groups: the Helfer Skin Tap technique group, the ShotBlocker technique group, and the control group (standard intramuscular injection). The effectiveness of non-pharmacological pain management techniques in reducing dysmenorrhea pain will be compared across these groups.
Masking Description: "In this study, both the participants and the investigators are aware of the intervention being applied. Participants in the Helfer Skin Tap Technique (HSTT) group, ShotBlocker group, and control group are informed about the specific treatment they receive."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Helfer Skin Tap Technique Group (Experimental): This group will receive the Helfer Skin Tap Technique (HSTT) as a non-pharmacological pain management intervention during intramuscular injection for dysmenorrhea. The effectiveness of this technique in reducing pain will be evaluated.
  Interventions: Behavioral: Halfer Skin Tape Technique
- 2.ShotBlocker Technique Group (Experimental): This group will receive the ShotBlocker technique during intramuscular injection for dysmenorrhea as a non-pharmacological pain management intervention. The effectiveness of this technique in reducing pain will be evaluated.
  Interventions: Behavioral: ShotBlocker Technique
- 3. Control Group (Placebo Comparator): This group will receive a standard intramuscular injection (IM) without any additional pain management technique. The pain intensity in this group will be compared to the other intervention groups.
  Interventions: Other: Standard Intramusculer injection

INTERVENTIONS:
Behavioral: Halfer Skin Tape Technique — Helfer Skin Tap Technique (HSTT) is a non-pharmacological pain management method that involves a series of gentle taps on the skin prior to an intramuscular injection. This technique is intended to distract the patient from the pain of the injection and reduce perceived pain intensity by stimulating different sensory pathways.
  Arms: 1. Helfer Skin Tap Technique Group
Behavioral: ShotBlocker Technique — ShotBlocker is a non-pharmacological device that applies pressure to the skin at the injection site to disrupt pain signals and reduce the pain perception during intramuscular injections. The pressure stimulates the sensory nerve fibers, which helps block the sharp pain from the needle insertion.
  Arms: 2.ShotBlocker Technique Group
Other: Standard Intramusculer injection — The control group will receive a standard intramuscular injection without the use of any pain management techniques (such as HSTT or ShotBlocker). This group serves as a baseline to compare the effect
  Arms: 3. Control Group

SUMMARY:
Brief Summary:

This study investigates the effectiveness of non-pharmacological techniques for managing dysmenorrhea (menstrual pain) in adolescents. The study focuses on methods such as Helfer Skin Tap Technique (HSTT) and ShotBlocker, which aim to reduce pain without medication. The goal is to determine how these techniques can help adolescents manage their pain more effectively.

The study targets adolescents aged 12-18 who experience menstrual pain. Participants will be monitored over several months to assess the impact of these techniques on their pain levels, emotional well-being, and daily activities.

Participation in the study poses minimal risks. However, the effectiveness of these pain management techniques may vary from person to person. By the end of the study, the aim is to improve pain management strategies for adolescents and gain a better understanding of the effectiveness of non-pharmacological treatments for dysmenorrhea.

DETAILED DESCRIPTION:
Objective:

The purpose of this study is to evaluate the effectiveness of non-pharmacological pain management techniques, namely the Helfer Skin Tap Technique (HSTT) and ShotBlocker, in reducing pain intensity during intramuscular injections in adolescents who present with dysmenorrhea (menstrual pain) in the emergency department. This study compares these techniques with a control group receiving standard intramuscular (IM) injection procedures.

Study Design:

This is a randomized controlled trial (RCT) designed to assess the pain-reducing effects of two non-pharmacological techniques during intramuscular injections. The study took place at Ladik State Hospital Emergency Department from October 1, 2025, to April 1, 2025. Participants were adolescent girls aged 12-18 years presenting to the emergency department with dysmenorrhea. The study compares the following groups:

* Group 1: Participants who receive Helfer Skin Tap Technique (HSTT).
* Group 2: Participants who use the ShotBlocker device.
* Control Group: Participants who receive standard intramuscular injection without any pain management techniques.

Hypotheses:

1. First Hypothesis (H₁): The group receiving Helfer Skin Tap Technique (HSTT) will experience lower pain intensity during the intramuscular injection compared to the group receiving the ShotBlocker technique and the control group.
2. Second Hypothesis (H₂): The group using the ShotBlocker will experience lower pain intensity during the intramuscular injection compared to the control group.
3. Third Hypothesis (H₃): The group receiving Helfer Skin Tap Technique (HSTT) will experience lower pain intensity compared to the group using the ShotBlocker technique.
4. Fourth Hypothesis (H₄): The control group will experience higher pain intensity compared to the groups receiving Helfer Skin Tap Technique (HSTT) or ShotBlocker.

Study Procedure:

Adolescents aged 12-18 years experiencing dysmenorrhea were randomly assigned to one of three groups: Helfer Skin Tap Technique (HSTT), ShotBlocker, or the control group. The pain intensity during the intramuscular injection was assessed using the Visual Analog Scale (VAS), a widely used method for measuring pain intensity. Pain ratings were recorded immediately after the injection, and follow-up evaluations were conducted to assess the continued effects on pain and emotional well-being.

Expected Outcomes:

We anticipate that both the Helfer Skin Tap Technique and ShotBlocker will reduce pain intensity during the injection, with the Helfer Skin Tap Technique (HSTT) potentially offering the most significant reduction in pain compared to the ShotBlocker and the control group. Secondary outcomes include emotional well-being, quality of life related to menstrual pain, and any adverse events related to the techniques used.

Risk and Safety Considerations:

The risks associated with participation in this study are minimal. The primary risk is mild discomfort or temporary soreness from the techniques being applied, which is rare and usually resolves quickly. All participants will be monitored for any adverse effects during the study. The techniques used, including HSTT and ShotBlocker, are safe, non-invasive, and commonly used in clinical settings.

Data Collection and Analysis:

Pain levels will be measured using the Visual Analog Scale (VAS), and data will be statistically analyzed to compare the effectiveness of each technique. We will evaluate the difference in pain intensity between the three groups and assess the feasibility of these non-pharmacological techniques for managing dysmenorrhea in adolescent girls. Statistical methods, including ANOVA and t-tests, will be employed to analyze the data.

Conclusion:

This study aims to provide evidence on the effectiveness of non-pharmacological pain management techniques, specifically the Helfer Skin Tap Technique (HSTT) and ShotBlocker, in reducing pain intensity in adolescents with dysmenorrhea during intramuscular injections. If successful, the findings could lead to better pain management options for adolescents, offering them drug-free solutions for managing menstrual pain, thus improving their quality of life.

ELIGIBILITY:
nclusion Criteria:

* Adolescents aged 12-18 years.
* Experience of dysmenorrhea (menstrual pain) during at least one menstrual cycle.
* Adolescents presenting to the emergency department with dysmenorrhea.
* Written informed consent from participants or their legal guardians.

Exclusion Criteria:

* Individuals with severe cardiovascular, neurological, or other serious medical conditions.
* Pregnant individuals.
* Individuals undergoing regular hormonal therapy or using birth control methods.
* Individuals with significant psychological or physiological conditions related to pain sensitivity (e.g., hyperalgesia).
* Individuals receiving other pharmacological treatments or pain management medications during the study.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Pain Perceived During Injection Using Helfer Skin Tap and ShotBlocker Techniques | within 5 minutes post-injection, 10 minutes, 30 minutes
  Reduction in Pain Intensity During Injection Using Helfer Skin Tap and ShotBlocker Techniques Pain intensity will be measured immediately after the intramuscular injection using the Visual Analog Scale (VAS), which ranges from 0 ("no pain") to 10 ("worst pain imaginable").

CONTACTS AND LOCATIONS:
Locations (1):
- Ladik Devlet Hastanesi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
"IPD will not be shared due to privacy and confidentiality concerns. All participant data will be anonymized and kept confidential in accordance with ethical guidelines and institutional review board (IRB) requirements. Additionally, there are no plans to share the data with other researchers as it is not necessary for the goals of this study."

REFERENCES:
- See also: This study was conducted to evaluate the effects of ShotBlocker and Palm Stimulator, developed by researchers, on reducing pain during intramuscular injections in 7-10 years old children.Material and Method: The study was conducted with three groups usin — https://acikbilim.yok.gov.tr/handle/20.500.12812/122468
- See also: The Effect of Buzzy Method on Reducing Pain During Intramuscular Injection in Children. Hasan Kalyoncu University, Graduate Education Institute, Department of Nursing, Master Thesis, Gaziantep, 2022. There search was carried out as a randomized controlle — https://tez.yok.gov.tr/UlusalTezMerkezi/TezGoster?key=kScA8XnrRb0WogX-qPGFkskAxpWgS7oPxXLAO7Y8emdlrs8idIHyUX6qoF4dV_El
- See also: The effects of vibration and pressure methods on the level of fear, anxiety, and pain of pediatric patients who were admitted to the emergency department for intramuscular injection were evaluated. — https://pubmed.ncbi.nlm.nih.gov/38171061/
- See also: The study purpose was to determine the decrease of dysmenorrhea pain rate after being given abdominal stretching exercise on nursing students at STIKES TanawaliPersada, Takalar, Indonesia. — https://iopscience.iop.org/article/10.1088/1742-6596/1028/1/012103